CLINICAL TRIAL: NCT00292097
Title: A Prospective, Randomized Trial of Early Versus Conventional Conversion From Endotracheal Intubation to Percutaneous Tracheostomy for Ventilatory Support of Trauma Patients With Severe Brain Injury
Brief Title: A Prospective, Randomized Trial of Early Versus Late Tracheostomy in Trauma Patients With Severe Brain Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty obtaining enrollment
Sponsor: Memorial Medical Center (Other)
Responsible Party: Russel Dumire, MD, FACS/MMC Progeam Director, General Surgery Residency Program, Memorial Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMC 05-27
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2008-06-05 (Estimated); Status verified 2008-06

CONDITIONS: Respiratory Failure; Traumatic Brain Injury
Keywords: Respiratory failure; Tracheostomy; Percutaneous dilatation tracheostomy; Endotracheal Conversion; Traumatic brain injury
MeSH Terms: conditions — Respiratory Insufficiency; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Early conversion from endotracheal intubation to percutaneous tracheostomy for ventilator support of trauma patients with severe brain injury
  Interventions: Procedure: Early tracheostomy
- 2 (Active Comparator): Conventional conversion from endotracheal intubation to percutaneous tracheostomy for ventilator support of trauma patients with severe brain injury
  Interventions: Procedure: Late tracheostomy

INTERVENTIONS:
Procedure: Early tracheostomy — early conversion - less than or equal to 72 hours
  Arms: 1
Procedure: Late tracheostomy — Late conversion (10-14 days)
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy of early conversion tracheostomy from endotracheal intubation (ET) to percutaneous, dilatational tracheostomy (PDT) in traumatic brain-injured patients requiring prolonged mechanical ventilation.

DETAILED DESCRIPTION:
This is a prospective, randomized trial to evaluate the efficacy of early (less than or equal to 72 hours) versus late (10 to 14 days) conversion from endotracheal intubation to percutaneous, dilatational, translaryngeal tracheostomy for mechanical ventilation of traumatic brain injured patients.

The primary efficacy parameter will be the number of days on mechanical ventilation.

Secondary objectives include:

* Number of days in the hospital
* To assess the incidence of ventilator-acquired pneumonia in each group
* To assess the incidence of accidental extubation in each group
* To assess the incidence of death in each group

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* TBI defined as penetrating or blunt brain injury including 1)subarachnoid hemorrhage, 2)subdural hemorrhage, 3) epidural hemorrhage, 4)brain contusion, 5)diffuse axonal injury
* mechanically ventilated by endotracheal intubation
* projected to need ventilation support for more than 14 days according to: GCS measured in field less than or equal to 8 and a GCS on day 3 which remains less than or equal to 8
* informed consent obtained from patient or legal representative

Exclusion Criteria:

* less than 18 years of age
* projected to need ventilation support for less than 14 days
* anatomical deformity of the neck, including thyromegaly and cervical tumors
* previous tracheostomy
* uncontrolled coagulopathy
* existence of platelet count less than 50,000/mm2
* anti-platelet agents
* clinical evidence of ongoing infection at the proposed tracheostomy site as per physician
* mechanical ventilation with a positive end-expiratory pressure greater than 12 cm H20
* intubated more than 72 hours
* patient has undergone cricothyroidotomy
* cricoid cartilage, trachea, or sternal notch not palpable with neck in position

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Total number of mechanical ventilation days | until discharged

SECONDARY OUTCOMES:
Total number of hospital days | until discharged
Incidence of ventilator-associated pneumonia | until discharged
Incidence of accidental extubation | until discharged
Incidence of death | until discharged

CONTACTS AND LOCATIONS:
Overall Officials: Russell D Dumire, MD, Principal Investigator — Memorial Medical Center; Stephen L Miller, MD, Principal Investigator — Memorial Medical Center
Locations (1):
- Memorial Medical Center, Johnstown, Pennsylvania, United States